CLINICAL TRIAL: NCT03137173
Title: A Randomized, Double-blind, Multicenter Study to Establish the Safety and Efficacy of Ceftobiprole Medocaril Compared With Vancomycin Plus Aztreonam in the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Ceftobiprole in the Treatment of Patients With Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPR-CS-008
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — ceftobiprole medocaril; ceftobiprole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ceftobiprole medocaril (Experimental): Patients treated with ceftobiprole medocaril 500 mg q8h (with dose adjustment for renal impairment).
  Interventions: Drug: ceftobiprole medocaril
- vancomycin+aztreonam (Active Comparator): Patients treated with vancomycin 1000 mg (or 15 mg/kg) q12h plus aztreonam 1000 mg q12h (both with dose adjustment for renal impairment).
  Interventions: Drug: vancomycin+aztreonam

INTERVENTIONS:
Drug: ceftobiprole medocaril — ceftobiprole 500 mg was to be administered every 8 hours as a 2-hour IV infusion (with dose adjustment for renal impairment). The treatment duration was for a minimum of 5 days and a maximum of 10 days. Treatment could be extended up to 14 days if in the investigator's opinion this was required, and the extension was approved by the sponsor's medical monitor.
  Other Names: ceftobiprole
  Arms: ceftobiprole medocaril
Drug: vancomycin+aztreonam — Vancomycin 1000 mg (or 15 mg/kg) was to be administered every 12 hours (with dose adjustment for renal impairment) as 2-hour IV infusion. Vancomycin dose adjustment for morbidly obese and hypermetabolic patients was to be done according to local standard of care. When locally available, vancomycin trough testing (VTT) might have been used by the unblinded pharmacist or delegate to adjust the vancomycin dose. The treatment duration was for a minimum of 5 days and a maximum of 10 days. Treatment could be extended up to 14 days if in the investigator's opinion this was required, and the extension was approved by the sponsor's medical monitor.
  Aztreonam 1000 mg was to be administered as a 0.5-hour IV infusion every 12 hours. If CLCR was < 30 mL/min (i.e., severe renal impairment), the aztreonam dosage regimen was to be adjusted. The requirement to continue aztreonam therapy beyond Day 3 was to be reassessed at the 72-hour study visit.
  Arms: vancomycin+aztreonam

SUMMARY:
This was a randomized, double-blind, active-controlled, parallel-group, multicenter study in adult hospitalized patients to establish the safety and efficacy of ceftobiprole medocaril compared with vancomycin plus aztreonam in the treatment of acute bacterial skin and skin structure infections (ABSSSIs).

DETAILED DESCRIPTION:
This was a randomized, double-blind, active-controlled, parallel-group, multicenter study in adult hospitalized patients with ABSSSIs. Randomization was stratified by study site and type of ABSSSI (with major cutaneous abscess comprising ≤ 30% of the Intent-to-Treat [ITT] population).

Primary endpoint for FDA: Early clinical response based on the percent reduction in lesion size at 48-72 hours compared to baseline in patients who did not receive rescue therapy and were alive, in the ITT population.

Primary endpoint for EMA: Investigator-assessed clinical success at the test-of-cure (TOC) visit 15-22 days after randomization, in the co-primary ITT and Clinically Evaluable (CE) populations.

ELIGIBILITY:
INCLUSION CRITERIA

1. Male or female, aged ≥18 years.
2. Diagnosis of ABSSSI, meeting at least one of the definitions in (a) to (c) below. Local symptoms must have started within the 7 days prior to the Screening visit:

   1. Cellulitis/erysipelas, defined as a diffuse skin infection characterized by all of the following within 24 hours:

      * i. Rapidly spreading areas of erythema, edema, and/or induration with a minimum total lesion surface area of 75cm^2
      * ii. No collection of pus apparent upon visual examination
      * iii. At least two of the following local signs of infection:

        * erythema
        * induration
        * localized warmth
        * pain or tenderness on palpation
        * swelling/edema
   2. Major cutaneous abscess, defined as infection characterized by a collection of pus within the dermis or deeper that is apparent upon visual examination before or after therapeutic intervention and is accompanied by all of the following within 24 hours:

      * i. Erythema, edema and/or induration with a minimum total lesion surface area of 75 cm^2.
      * ii. At least two of the following local signs of infection:

        * fluctuance
        * incision and drainage required
        * purulent or seropurulent drainage
        * localized warmth
        * pain or tenderness on palpation
   3. Wound infection, defined as infection of any apparent break in the skin characterized by at least one of the following:

      * i. Superficial incision/surgical site infection meeting all of the following criteria:

        * involves only the skin or subcutaneous tissue around the incision (does not involve fascia).
        * occurs within 30 days of procedure.
        * purulent drainage (spontaneous or therapeutic) with surrounding erythema, edema and/ or induration with a minimum total lesion surface area of 75cm^2.
      * ii. Post-traumatic wound (including penetrating trauma, e.g., needle, nail, knife, insect and spider bites) meeting the following criterion within 24 hours:

        * Purulent drainage (spontaneous or therapeutic) with surrounding erythema, edema and/or induration with a minimum total lesion surface area of 75cm^2.
3. At least one of the following regional or systemic signs of infection at the Screening visit:

   1. Lymph node tenderness and volume increase, or palpable lymph node proximal to the primary ABSSSI.
   2. Fever > 38 °C/100.4 °F measured orally, > 38.5 °C / 101.3 °F measured tympanically, > 37.5 °C / 99.5 °F measured by the axillary method, or > 39 °C / 102.2 °F measured rectally.
   3. White blood cell (WBC) count > 10.0 × 10^9/L or < 4.0 × 10^9/L.
   4. > 10% immature neutrophils (band forms).
4. Requirement for IV antibacterial treatment.
5. Willing and able to adhere to study procedures (including prohibitions and restrictions) as specified in this protocol.
6. Willing and able to remain hospitalized (in a hospital or equivalent medical confinement or clinical research unit) until completion of the early-clinical-response assessment for the primary endpoint.
7. Informed consent signed by the patient, or their legally acceptable representative if appropriate, indicating that they understand the purpose of, and procedures required for, the study, and are willing to participate.

EXCLUSION CRITERIA

Patients meeting any one of the following:

1. Use of any systemic antibacterial treatment within 14 days, or topical antibacterial administration on the primary lesion within 96 hours, before first infusion of study drug.

   Exception: Receipt of a single dose of a short acting (half-life ≤ 12 hours) antibacterial therapy (e.g., for surgical prophylaxis) within > 3 days before randomization (i.e., patients cannot have received any antibacterial treatment within 72 hours of randomization).
2. Contraindication to the administration of either of the study treatments, including known clinically-relevant hypersensitivity to related antibacterial treatments (e.g., beta-lactam and glycopeptide antibiotics), or to metronidazole if required as adjunctive therapy.
3. Participation in any other clinical study within the 30 days prior to randomization, or any prior participation in this study.
4. The primary ABSSSI is an uncomplicated skin and skin structure infection, such as furuncles, minor abscesses (area of suppuration not surrounded by cellulitis/erysipelas), impetiginous lesions, superficial or limited cellulitis/erysipelas, or minor wound infections (e.g., stitch abscesses).
5. The primary ABSSSI is due to, or associated with, any of the following:

   1. Diabetic foot infection, gangrene, or perianal abscess.
   2. Concomitant infection at another site (e.g., septic arthritis, endocarditis, osteomyelitis), not including a secondary ABSSSI lesion.
   3. Infected burns.
   4. Decubitus or chronic skin ulcer, or ischemic ulcer due to peripheral vascular disease (arterial or venous).
   5. Any evolving necrotizing process (e.g., necrotizing fasciitis).
   6. Infections at vascular catheter sites, or involving thrombophlebitis.
6. The primary ABSSSI is associated with, or in close proximity to, a prosthetic device.
7. Patients who are placed in a hyperbaric chamber as adjunctive therapy for the ABSSSI.
8. Patients expected to require more than two surgical interventions in the operating room for the ABSSSI.
9. Severe sepsis or septic shock.
10. Significant or life-threatening condition (e.g., endocarditis, meningitis) that would confound, or interfere with, the assessment of the ABSSSI.
11. Another severe, acute or chronic medical condition, psychiatric condition, or laboratory abnormality that may increase the risks associated with study participation or administration of the investigational product, or may interfere with the interpretation of study results, and which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Receiving treatment for active tuberculosis.
13. Absolute neutrophil count < 0.5 × 10^9/L.
14. Recent history of opportunistic infections (i.e., within 30 days) if the underlying cause of these infections is still active (e.g., leukemia, transplant, acquired immunodeficiency syndrome [AIDS]).
15. Patients receiving systemic steroids (> 40 mg per day prednisolone, or equivalent), or receiving immunosuppressant drugs.
16. Requirement for peritoneal dialysis, plasmapheresis, hemodialysis, venovenous dialysis, or other forms of renal filtration, or expected to require such treatment before the TOC visit.
17. Alanine transaminase (ALT) or aspartate transaminase (AST) levels ≥ 8× the upper limit of normal, OR severe hepatic disease with Child-Pugh class C.
18. Women who are pregnant or nursing.
19. Women who are of childbearing potential and unwilling to use an acceptable method of birth control during the study: female sterilization (bilateral tubal occlusion or oophorectomy, or hysterectomy) or male partner vasectomy; intrauterine device (IUD); combined (estrogen and progesterone containing) hormonal contraception (oral, vaginal ring, or transdermal patch) with an ethinylestradiol dose of at least 30 µg, plus use of male condoms (preferably with spermicides), female condoms, a female diaphragm or a cervical cap; or total sexual abstinence.

    Women are not considered to be of childbearing potential if they are either ≥ 1 year post-menopausal (where menopause is defined as at least 12 months of amenorrhea), or have a serum follicle stimulating hormone (FSH) measurement consistent with post-menopausal status according to local laboratory thresholds. An FSH measurement at Screening is to be obtained for post-menopausal females aged < 50 years, or for those aged ≥ 50 years who have been post-menopausal for < 2 years.
20. Inability to start study-drug therapy within 24 hours of Screening.
21. Patients with illicit drug use within 12 months of screening, including heroin, other opioids (unless prescribed for medical reasons unrelated to heroin substitution), cocaine / crack cocaine, and amphetamine or methamphetamine. Exception: Cannabis use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica
Locations (34):
- United States (16):
  - Physician Alliance Research Center, Anaheim, California
  - Saint Joseph's Clinical Research, Anaheim, California
  - eStudySite - Chula Vista - PPDS, Chula Vista, California
  - Central Valley Research LLC, Fresno, California
  - Marvel Clinical Research, Huntington Beach, California
  - eStudySite - La Mesa - PPDS, La Mesa, California
  - Omnibus Clinical Research, La Palma, California
  - Alliance Research LLC, Long Beach, California
  - Long Beach Clinical Trials, Long Beach, California
  - Central Valley Research, LLC, Modesto, California
  - Gonzalez MD and Aswad MD Health Services, Coral Gables, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Mercury Street Medical Group, Butte, Montana
  - eStudySite - Las Vegas - PPDS, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment, Pleven
  - University Multiprofile Hospital for Active Treatment, Plovdiv
  - University Multiprofile Hospital for Active Treatment, Rousse
  - "University Multiprofile Hospital for Active Treatment and Emergency Medicine ""N. I. Pirogov"", Clinic of Purulent-Septic Surgery-"N.I. Pirogov"", Sofia
- Hungary (4):
  - Kaposi Mor Teaching Hospital, Kaposvár
  - CRU Hungary Ltd., Miskolc
  - University of SzegednAlbert Szent-Gyorgyi Clinical Center, Szeged
  - Csolnoky Ferenc Hospital, Veszprém
- Ukraine (10):
  - Dnipropetrovsk I.I. Mechnуkov Regional Clinical Hospital, Surgery Department #2, Dnipro
  - Ivano-Frankivsk City Clinical Hospital Surgery 1, Ivano-Frankivsk
  - Ivano-Frankivsk City Clinical Hospital General Surgery, Ivano-Frankivsk
  - Kyiv City Clinical Hospital, Kyiv
  - Public City Clinical Hospital of Emergency Medical Care, Lviv
  - Lviv Regional Clinical Hospital, Lviv
  - Central City Clinical Hospital, Uzhhorod
  - Vinnytsia M.I. Pyrohov Regional Clinical Hospital, Vinnytsia
  - Zaporizhia City Clinical Hospital of Urgent and Emergency Medical Care, Zaporizhia
  - Central District Hospital, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welte T, Scheeren TW, Overcash JS, Saulay M, Engelhardt M, Hamed K. Efficacy and safety of ceftobiprole in patients aged 65 years or older: a post hoc analysis of three Phase III studies. Future Microbiol. 2021 May;16:543-555. doi: 10.2217/fmb-2021-0042. Epub 2021 May 7. PMID 33960817
- [Derived] Overcash JS, Kim C, Keech R, Gumenchuk I, Ninov B, Gonzalez-Rojas Y, Waters M, Simeonov S, Engelhardt M, Saulay M, Ionescu D, Smart JI, Jones ME, Hamed KA. Ceftobiprole Compared With Vancomycin Plus Aztreonam in the Treatment of Acute Bacterial Skin and Skin Structure Infections: Results of a Phase 3, Randomized, Double-blind Trial (TARGET). Clin Infect Dis. 2021 Oct 5;73(7):e1507-e1517. doi: 10.1093/cid/ciaa974. PMID 32897367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with an ABSSSI who received any systemic antibacterial treatment within 14 days, or topical antibacterial administration on the primary lesion within 96 hours, before first infusion of study drug were not allowed to enter the study. Hospitalization in a medical clinic was mandatory for the first 72 hours.
Pre-assignment Details: 3 randomized patients were not dosed, due to ICF withdrawal (2 patients) and death (1 patient).
Groups:
- Ceftobiprole Medocaril: Patients treated with ceftobiprole medocaril 500 mg every 8 hours (with dose adjustment for renal impairment).
- Vancomycin+Aztreonam: Patients treated with vancomycin 1000 mg (or 15 mg/kg) every 12 hours plus aztreonam 1000 mg every 12 hours (both with dose adjustment for renal impairment). Vancomycin dose adjustment for obese and hypermetabolic patients was according to local standard of care. The requirement for aztreonam therapy was to be reassessed at the 72-hour study visit.
Period: Overall Study
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam
Started | 335 | 344
Completed | 309 | 308
Not Completed | 26 | 36
Not completed — Withdrawal by Subject | 8 | 13
Not completed — Death | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 13 | 18
Not completed — Other reasons | 3 | 2

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Ceftobiprole Medocaril: Patients treated with ceftobiprole medocaril 500 mg every 8 hours (with dose adjustment for renal impairment). Duration of infusion: 2 hours.
- Vancomycin+Aztreonam: Vancomycin 1000 mg (or 15 mg/kg) every 12 hours plus aztreonam 1000 mg every 12 hours (both with dose adjustment for renal impairment). Vancomycin dose adjustment for obese and hypermetabolic patients was according to local standard of care. The requirement for aztreonam therapy was to be reassessed at the 72-hour study visit. Duration of vancomycin infusion: 2 hours; duration of aztreonam infusion: 0.5 hours.
- Total: Total of all reporting groups
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam | Total
Number analyzed (Participants) | 335 | 344 | 679
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 294 | 292 | 586
  >=65 years | 41 | 52 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 143 | 280
  Male | 198 | 201 | 399
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 318 | 330 | 648
  Black or African American | 7 | 8 | 15
  Asian | 0 | 1 | 1
  American Indian or Alaska Native | 4 | 3 | 7
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 5 | 2 | 7
  Hispanic or Latino | 103 | 115 | 218
Region of Enrollment [Number; unit: participants]
  Hungary | 2 | 1 | 3
  United States | 203 | 215 | 418
  Ukraine | 82 | 80 | 162
  Bulgaria | 48 | 48 | 96
Type of ABSSSI [Count of Participants; unit: Participants]
  Cellulitis/erysipelas | 112 | 111 | 223
  Major cutaneous abscess | 96 | 93 | 189
  Wound infection | 127 | 140 | 267

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response
Description: Comparison of early clinical response, including ≥ 20% reduction from baseline in the primary lesion area (based on ruler measurements), survival for ≥ 72 hours and no rescue therapy in the ITT population
Time Frame: 48-72 hours after start of study drug treatment
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam
Number analyzed (Participants) | 335 | 344
Participants | 306 | 303
Statistical Analysis 1: Comparison: Ceftobiprole Medocaril vs Vancomycin+Aztreonam; Test type: Non-Inferiority — Non-inferiority was assessed by the two-sided 95% confidence interval (CI) of the between-group difference (ceftobiprole minus vancomycin+aztreonam) using a 10% non-inferiority margin in the ITT population. Difference was computed using the Cochran-Mantel-Haenszel (CMH) weights method, adjusted for geographical region and actual type of ABSSSI; Risk Difference (RD) = 3.3, 95% CI 2-sided [-1.2 to 7.8]

2. Secondary Outcome: Investigator-assessed Clinical Success in the ITT Population
Description: Comparison of investigator-assessed clinical success (based on resolution of baseline signs and symptoms of the primary infection) in the ITT population
Time Frame: 15-22 days after randomization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam
Number analyzed (Participants) | 335 | 344
Participants | 302 | 306
Statistical Analysis 1: Comparison: Ceftobiprole Medocaril vs Vancomycin+Aztreonam; Test type: Non-Inferiority — Non-inferiority was assessed by the two-sided 95% CI of the between-group difference (ceftobiprole minus vancomycin+aztreonam) using a 10% non-inferiority margin in the ITT population. Difference was computed using the CMH weights method, adjusted for geographical region and actual type of ABSSSI; Risk Difference (RD) = 1, 95% CI 2-sided [-3.5 to 5.6]

3. Secondary Outcome: Investigator-assessed Clinical Success in the Clinically Evaluable (CE) Population
Description: Comparison of investigator-assessed clinical success (based on resolution of baseline signs and symptoms of the primary infection) in the clinically evaluable (CE) population
Time Frame: 15-22 days after randomization
Population: CE population
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam
Number analyzed (Participants) | 283 | 293
Participants | 277 | 279
Statistical Analysis 1: Comparison: Ceftobiprole Medocaril vs Vancomycin+Aztreonam; Test type: Non-Inferiority — Non-inferiority was assessed by the two-sided 95% CI of the between-group difference (ceftobiprole minus vancomycin plus aztreonam) using a 10% non-inferiority margin in the CE populations. Difference was computed using the CMH weights method, adjusted for geographical region and actual type of ABSSSI; Risk Difference (RD) = 2.7, 95% CI 2-sided [-0.3 to 5.6]

ADVERSE EVENTS:
Time Frame: Up to 35 days after last treatment
Groups:
- Ceftobiprole Medocaril: Patients treated with ceftobiprole medocaril 500 mg every 8 hours (with dose adjustment for renal impairment).
  Ceftobiprole medocaril: A reconstituted solution of 500 mg of ceftobiprole in 250 mL of water for injection was administered IV every 8 hours (with dose adjustment for renal impairment) for a minimum of 5 days and a maximum of 10 days. Treatment could be extended up to 14 days if in the investigator's opinion this was required, and the extension was approved by the sponsor's medical monitor. Duration of each infusion: 2 hours.
- Vancomycin+Aztreonam: Patients treated with vancomycin 1000 mg (or 15 mg/kg) every 12 hours plus aztreonam 1000 mg every 12 hours (both with dose adjustment for renal impairment).
  Vancomycin+aztreonam: vancomycin 1000 mg (or 15 mg/kg) every 12 hours (with dose adjustment for renal impairment). Vancomycin dose adjustment for obese and hypermetabolic patients was according to local standard of care. Duration of infusion: 2 hours.
  Aztreonam for Injection for IV infusion must have been reconstituted with at least 3 mL sterile water for injection. The reconstituted solution of aztreonam must have been further diluted with 100 mL NaCl 0.9% solution for injection, resulting in an aztreonam concentration of 10 mg/mL (1%). Aztreonam 1000 mg was to be administered as a 0.5-hour IV infusion every 12 hours. If CLCR was < 30 mL/min (i.e., severe renal impairment), the aztreonam dosage regimen might have been adjusted. The requirement for aztreonam therapy was to be reassessed at the 72-hour study visit.
Arm/Group | Ceftobiprole Medocaril | Vancomycin+Aztreonam
All-Cause Mortality (participants affected / at risk) | 1/334 | 3/342
Serious Adverse Events (participants affected / at risk) | 6/334 | 12/342
Other Adverse Events (participants affected / at risk) | 63/334 | 47/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole Medocaril (N=334) | Vancomycin+Aztreonam (N=342)
CARDIAC ARREST (Cardiac disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 1
MULTIPLE ALLERGIES (Immune system disorders) | 0 | 1
SKIN BACTERIAL INFECTION (Infections and infestations) | 1 | 3
CELLULITIS (Infections and infestations) | 0 | 2
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole Medocaril (N=334) | Vancomycin+Aztreonam (N=342)
Nausea (Gastrointestinal disorders) | 36 | 20
Diarrhoea (Gastrointestinal disorders) | 21 | 16
Headache (Nervous system disorders) | 19 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03137173/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03137173/SAP_001.pdf